CLINICAL TRIAL: NCT00180791
Title: Treatment Protocol for High-Risk PNET Brain Tumors in Children With Surgery, Sequential Chemotherapy, Conventional and High-Dose With Peripheral Blood Stem Cell Transplantation and Radiation Therapy
Brief Title: High Risk Primitive Neuroectodermal (PNET) Brain Tumors in Childhood
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNET HR
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2006-09

CONDITIONS: Medulloblastoma; Brain Tumors; Neuroectodermal Tumors, Primitive
Keywords: Brain PNET
MeSH Terms: conditions — Medulloblastoma; Brain Neoplasms; Neuroectodermal Tumors, Primitive | interventions — Etoposide; Carboplatin; Melphalan; Cisplatin; Thiotepa

INTERVENTIONS:
Drug: Etoposide, carboplatin, melphalan, cisplatin, thiotepa

SUMMARY:
The purpose of this study is to evaluate the efficacy of the combination of surgery, conventional chemotherapy, sequential high-dose chemotherapy with peripheral blood stem cell transplantation and reduced dose radiation therapy in high-risk PNET brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Medulloblastoma in patients less than 5 years of age
* Brain PNET in patients less than 10 years of age
* Histologically documented diagnosis
* Body weight of > 8 kg

Exclusion Criteria:

* Parents' refusal

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Estimated)
Dates: Start 2002-07

PRIMARY OUTCOMES:
Response of medulloblastoma metastases to the chemotherapy regimen in children less than 5 years of age
Progression-free survival of children less than 10 years of age with brain PNET

SECONDARY OUTCOMES:
Progression-free survival of children less than 5 years of age with metastatic medulloblastoma
Toxicity
Long term sequelae

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Kalifa, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France